CLINICAL TRIAL: NCT00375843
Title: Response Variability in Treatment Resistant Depression - an Ancillary Study to "Sequenced Treatment Alternatives to Relieve Depression (STAR*D)"
Brief Title: Brain Activity Changes and Treatment Response in Depressed People Who Are Receiving Antidepressant Medication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Ian A. Cook, MD, PI, University of California, Los Angelos
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH069217 (NIH); DATR A5-ETMA; R01 MH069180 (Alpert)
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2008-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram; Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Level 1 Treatment: Escitalopram (Active Comparator): Level 1 participants who are assigned to escitalopram
  Interventions: Drug: Escitalopram
- Level 2: Sertraline (Active Comparator): Participants from Level 1 who do not achieve remission with escitalopram enter Level 2 and switch to sertraline
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Escitalopram — Level 1 of the study involves open-label treatment with escitalopram, up to 30 mg/day for up to 12 weeks.
  Other Names: Lexapro
  Arms: Level 1 Treatment: Escitalopram
Drug: Sertraline — Level 2 of the study involves open-label treatment with sertraline, up to 200 mg/day for up to 12 weeks.
  Other Names: Zoloft
  Arms: Level 2: Sertraline

SUMMARY:
This study will examine how brain activity is affected by antidepressant treatment and how changes in brain activity relate to treatment response in people with depression.

DETAILED DESCRIPTION:
Depression is a serious medical illness that is characterized by a persistent sad, anxious, or empty mood. Many treatments have been shown to relieve depression, including both medications and behavioral therapies. No single treatment, however, works for everyone. Approximately half of the people being treated for depression do not respond to the first medication they try. Studies have shown that some people with depression show changes in brain activity within 2 weeks of starting treatment, even though symptoms do not change until later. People who do not respond to treatment, however, do not exhibit these changes in brain activity. More information is needed to understand the different ways in which people with depression respond to medication. This study will examine how brain activity is affected by antidepressant treatment and how changes in brain activity relate to treatment response in people with depression. It will also determine whether the brain testing involved in this study is burdensome to the participants.

Individuals interested in taking part in this 1-year study will first attend one screening visit to determine their eligibility for participation. Before beginning treatment, all participants will have an electroencephalogram (EEG) to determine baseline brain activity. Participants will then receive up to 12 weeks of treatment with escitalopram, an antidepressant medication. Study visits will be held every 2 to 3 weeks during this phase. At the Week 2 visit, participants will have another EEG. Participants who respond to escitalopram by the end of the treatment phase will be asked to participate in a 6-month follow-up phase, in which participants will be followed by their own personal physicians, but will have the option to continue treatment with escitalopram. Follow-up visits will be held at Months 3 and 6. Participants who do not respond to escitalopram by the end of the treatment phase will have another EEG, and will then receive up to 12 weeks of treatment with sertraline, another antidepressant medication. Study visits will be held every 2 to 3 weeks, and participants will have a fourth EEG at Week 2. Participants who respond to sertraline will then enter the 6-month follow-up phase, and may continue receiving sertraline. Participants who do not improve with sertraline will receive referrals for additional care outside of the study.

ELIGIBILITY:
Inclusion Criteria:

* Currently an outpatient with nonpsychotic, unipolar major depressive disorder (MDD)
* Score of 14 or greater on the 17-item Hamilton Rating Scale for Depression (HAM-D17)
* Antidepressant treatment is deemed appropriate by the study clinician
* Willing to use an effective form of contraception throughout the study

Exclusion Criteria:

* Mentally or legally incapacitated
* Lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder, MDD with psychotic features, or dementia
* Patients currently suffering from anorexia nervosa, bulimia nervosa, or obsessive compulsive disorder
* History of substance abuse disorder within 6 months prior to study entry
* Current suicidal ideation that would make outpatient treatment unsafe
* Past medication response that may make escitalopram or sertraline treatment unsafe or inappropriate (e.g., previous intolerance or lack of response to either medication)
* History of a failed treatment with escitalopram (40 mg or more) or sertraline (200 mg or more) during the current depressive episode
* Any medical conditions that would make treatment with escitalopram or sertraline medically inadvisable
* Unstable medical illness
* Unstable psychiatric illness likely to require inpatient treatment within the 6 months following study entry
* History of seizures, brain surgery, skull fracture, significant head trauma, or previous abnormal EEG
* Pregnant or plans to become pregnant within the 12 months following study entry
* Breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Relationship between depression symptoms and brain physiologic measures | Measured at exit from Level 1 treatment or from Level 2 treatment (each 12 weeks duration)

SECONDARY OUTCOMES:
Patient acceptability of EEG measures | Measured after final EEG recording
Relationship between brain physiologic measures and side effects | Measured at study exit
Relationship between brain physiologic measures and quality of life measures | Measured at study exit
Relationship between brain physiologic measures and psychosocial function measures | Measured at study exit
Relationship between brain physiologic measures and durability of remission, assessed as return of depressive symptoms during the 6 month follow-on phase | Measured at Month 6 of follow-on phase

CONTACTS AND LOCATIONS:
Overall Officials: Ian Cook, MD, Principal Investigator — UCLA Semel Institute
Locations (3):
- United States (3):
  - UCLA Semel Institute, Los Angeles, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Harvard/MGH, Boston, Massachusetts

REFERENCES:
- [Background] Leuchter AF, Cook IA, Witte EA, Morgan M, Abrams M. Changes in brain function of depressed subjects during treatment with placebo. Am J Psychiatry. 2002 Jan;159(1):122-9. doi: 10.1176/appi.ajp.159.1.122. PMID 11772700
- [Background] Cook IA, Leuchter AF, Morgan M, Witte E, Stubbeman WF, Abrams M, Rosenberg S, Uijtdehaage SH. Early changes in prefrontal activity characterize clinical responders to antidepressants. Neuropsychopharmacology. 2002 Jul;27(1):120-31. doi: 10.1016/S0893-133X(02)00294-4. PMID 12062912
- See also: Click here for the UCLA Depression Research website — http://www.DepressionResearch.com